CLINICAL TRIAL: NCT03604042
Title: Comparison of Two Regimens of Individualized, Adjustable Human Milk Fortification in Pretem Infants Using a New Modular Protein-only Fortifier
Brief Title: Comparison of Two Dose Adjustment Strategies of a Human Milk Protein Fortifier in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 13.01.INF
Record Dates: First submitted 2018-04-26; First posted 2018-07-27 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight-driven protein fortification (Active Comparator): Individualized protein fortification based on weight gain
  Interventions: Combination Product: Protein fortifier
- BUN-driven protein fortification (Experimental): Individualized protein fortification based on BUN concentrations
  Interventions: Combination Product: Protein fortifier

INTERVENTIONS:
Combination Product: Protein fortifier — Protein Fortifier to be added to Fortified human milk according to feeding regimen

SUMMARY:
The primary objective is to compare weight gain (g/day) of infants receiving new protein fortifier (PF) according to a blood urea nitrogen (BUN)-driven fortification regimen to weight gain (g/day) of infants receiving PF according to a weight-driven fortification regimen (standard of care) over a 21 day period.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age in weeks: 23 weeks 0 days and 31 weeks 6 days.
* Birth weight less or equal to 1500 g
* Minimum enteral intake of 150-160 mL/kg/d fortified HM
* Parents, liable parent, or legal representative (LR) if applicable are willing and able to sign written informed consent and written informed consent is obtained prior to trial entry

Exclusion Criteria:

* Infants with weight z-score < -2 SD, based on the Fenton growth chart (Fenton 2013)
* Intra-ventricular hemorrhage (grade 3-4) determined using cranial ultrasonography or periventricular leukomalacia.
* Renal disease determined by symptoms (oliguria, anuria, proteinuria, hematuria) associated with an increased creatinine.
* Cholestasis (total bilirubin > 5 mg/dL or 85 umol/L and direct bilirubin > 20% of total bilirubin) associated with one or more abnormal liver function tests (AST, ALT, or GGT).
* Major congenital malformations that may impact ability to accept enteral feedings (i.e., severe cleft palate, etc.).
* Suspected or documented systemic or congenital infections (i.e., human immunodeficiency virus, cytomegalovirus, etc.).
* Evidence of cardiac, respiratory, endocrinologic, hematologic, gastrointestinal, or other systemic diseases that may impact growth, e.g.,:

  * NEC grade above or equal to 2
  * Uncontrolled sepsis
* Suspected or documented maternal substance abuse:

  * Born to mothers who smoked > 10 cigarettes per day during pregnancy
  * Born to mothers who used illicit drugs (e.g. marijuana, cocaine, amphetamines, or heroin) or alcohol (> 3 alcoholic beverages per week) during pregnancy
* Subjects' parent(s) or legal representative who are not willing and not able to comply with scheduled visits and the requirements of the study protocol
* Infants who have received any experimental treatment or received any other investigational intervention (procedure or product) unrelated to this trial, prior to enrollment

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Comparison of weight gain | From Day 6 to Day 27
  To compare weight gain (g/day) of infants receiving new protein fortifier (PF) according to a BUN-driven fortification regimen to weight gain (g/day) of infants receiving PF according to a weight-driven fortification regimen

SECONDARY OUTCOMES:
Comparison of weight gain (g/day) of infants after 1 and 3 weeks of individualized protein fortification to weight gain during the 5-day period of standard Human Milk (HM) fortification | Day 6 to Day 13, and Day 6 to Day 27
  Comparison of weight gain (g/day) of infants after 1 and 3 weeks of individualized protein fortification to weight gain during the 5-day period of standard HM fortification
Changes in growth parameters: Lengths (crown-heel and knee-heel) and length gain (cm) | Day 6 to Day 27 (minimum)
  Changes in growth parameters: Lengths (crown-heel and knee-heel) and length gain (cm)
Changes in growth parameters: head circumference and head circumference gain (cm) | Day 6 to Day 27 (minimum)
  Changes in growth parameters: head circumference and head circumference gain (cm)
Changes in growth parameters: BMI and BMI changes (kg body weight/m^2) | Day 6 to Day 27 (minimum)
  Changes in growth parameters: BMI and BMI changes (kg body weight/m^2)
Body composition including lean fat mass and fat-free mass | Day 6 to Day 27 (minimum)
  Body composition including lean fat mass and fat-free mass
Weight at hospital discharge | Day 27 (minimum)
  Weight at hospital discharge
Macronutrient content in human milk | Day 6 to Day 27 (minimum)
  Macronutrient content in human milk using a Miris Human Milk Analyzer to measure the composition of the human milk
Feeding and gastrointestinal (GI) tolerance | Day 6 to Day 27 (minimum)
  Feeding and gastrointestinal (GI) tolerance determined using Digestive tolerance scores based on four binary parameters (0 = absence or 1 = presence) collected in daily routine care: Sore abdomen, liquid stools, gastric residuals, and regurgitation or vomiting
Safety evaluation including number of subjects with AEs | Day 1 to Day 27 (minimum)
  Safety evaluation including number of subjects with AEs
Biochemistry markers collected from blood and urine as part of routine NICU standard of care | Day 6 to Day 27 (minimum)
  Biochemistry markers collected from blood and urine as part of routine NICU standard of care: Routine biochemistries in Blood/Serum and Urine (in spot urine samples), and Nutrition markers in Blood/serum: albumin, pre-albumin, alkaline phosphatase, triglycerides and vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Paoli, Msc, Study Chair — Nestlé Research
Locations (1):
- Hopital de la Croix Rousse, Lyon, France